CLINICAL TRIAL: NCT06044259
Title: Randomized Trial on Acutely Dissected Aorta Repair With Hemiarch Replacement With or Without Stent Implantation (RADAR Trial)
Brief Title: Study Comparing Hemiarch Replacement and Hemiarch Plus Stent Implantation in Acute Aortic Dissection
Acronym: RADAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Randolph Wong, Professor and Chief of Division of Cardiothoracic Surgery, Department of Surgery, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE ref: 2023.075-T
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Aortic Dissection
Keywords: Hemiarch replacement; AMDS implantation
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Intervention Model Description: Randomized control trial of two groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hemiarch-AMDS (Active Comparator): Patient with acute DeBakey I aortic dissection will be put on GA and conventional CPB. During circulatory arrest, the aorta will be trimmed to the level of the distal ascending or proximal arch The AMDS device will be implanted into the aortic arch and descending thoracic aorta. The distal anastomosis will be done between a vascular graft and the distal ascending aorta/aortic arch including the AMDS device sewing cuff. After the distal anastomosis is completed, visceral and cerebral systemic perfusion and rewarming will be started. Proximal anastomosis will be performed and the patient will be weaned from cardiopulmonary bypass and decannulated.
  Interventions: Procedure: AMDS; Artivion, Atlanta, Georgia, US
- Hemiarch-C (Active Comparator): Patient with acute DeBakey I aortic dissection will be put on GA and conventional CPB. During circulatory arrest, the aorta will be trimmed to the level of the distal ascending or proximal arch The AMDS device will be implanted into the aortic arch and descending thoracic aorta. The distal anastomosis will be done between a vascular graft and the distal ascending aorta/aortic arch as per routine. After the distal anastomosis is completed, visceral and cerebral systemic perfusion and rewarming will be started. Proximal anastomosis will be performed and the patient will be weaned from cardiopulmonary bypass and decannulated.
  Interventions: Procedure: Conventional hemiarch replacement

INTERVENTIONS:
Procedure: AMDS; Artivion, Atlanta, Georgia, US — Ascyrus Medical Dissection Stent (AMDS; Artivion, Atlanta, Georgia, US) hybrid prosthesis which comprises a proximal sewing collar and a distal self-expanding nitinol un-covered stent.
  Arms: Hemiarch-AMDS
Procedure: Conventional hemiarch replacement — Coventional open hemiarch replacement
  Arms: Hemiarch-C

SUMMARY:
Acute DeBakey type I aortic dissection (ATAD) is one of the most lethal surgical emergencies. The conventional operative strategy is hemiarch replacement under cardiopulmonary bypass support to replace the diseased segment of the ascending aorta. However, in patients with dissection involving the whole aortic arch and descending thoracic aorta, the presence of the persistently perfused false lumen can lead to late aneurysm formation and require a second-stage operation, and this reduces long-term survival. In the surgical literature, there is growing evidence that the presence of Distal Anastomosis New Entry (DANE), which is a new intimal defect related to the trauma created by surgical sutures, is associated with persistent perfusion of the false lumen, aortic size growth, and the need of re-operation. The Ascyrus Medical Dissection Stent (AMDS; Artivion, Atlanta, Georgia, USA) is a hybrid prosthesis with a proximal sewing collar and distal nitinol self-expanding un-covered stent system designed to reduce the occurrence of DANE and hopefully depressurize the false lumen and lead to remodeling of the aortic wall.

The investigators plan to prospectively recruit consecutive patients with acute ascending thoracic aortic dissection patients (Excluding DeBakey II) and randomized them, after informed consent, into either the conventional hemiarch replacement group (Hemiarch-C) or the hemiarch replacement plus AMDS implantation group (Hemiarch-AMDS). The participating team will collect pre-operative, intra-operative and post-operative clinical and radiological parameters for two groups of patients. Written informed consent, specifically allowing the use of clinical records for this randomized study, will be obtained from every patient prior to data collection. Complete DICOM image files of the CT scans will be evaluated by two independent fully qualified Radiologists. Our primary outcome is the radiological detection of DANE in Hemiarch-C and Hemiarch-AMDS groups within the 12-month follow-up period.

This study will be the world's first randomized control trial in ATAD to compare the prevalence of DANE in Hemiarch-C and Hemiarch-AMDS. It could be a guideline-changing study for the treatment of ATAD and its impact on the immediate survival, second-stage treatment, and long-term survival of patients suffering from ATAD.

DETAILED DESCRIPTION:
Project Objectives

1. To compare the occurrence of Distal Anastomosis New Entry (DANE) after conventional hemiarch replacement group (Hemiarch-C) and the hemiarch replacement plus AMDS implantation group (Hemiarch-AMDS).
2. To compare the rate of all-cause mortality and aortic related mortality (at 30 days, 3-6, 12 months follow-up) between the study groups
3. To compare the rate of patients who are free from the following Major Adverse Events (MAEs) (new permanent disabling stroke, new permanent (> 30 days) paraplegia or paraparesis, reintervention, all-cause mortality) (at 12 months follow-up)
4. To compare radiological outcomes in terms of the rate of stenosis in supra-aortic head vessels, increasing (≥ 5 mm), stable or decreasing (≥ 5 mm) in true lumen in in both groups (at 3-6, 12 months follow-up).
5. To compare the radiological outcomes in terms of obliterated, completely thrombosed, partially thrombosed, or patent false lumen at various segments of aorta in both groups (at 3-6, 12 months follow-up).Thoracic aortic aneurysms (TAAs) and their complications (i.e. dissection, rupture, etc.) cause more than 1400 hospital admissions and 300 deaths every year in Hong Kong. Acute aortic dissection involving the ascending thoracic aorta is a highly lethal surgical emergency that warrants immediate surgical intervention. It can be classified according to DeBakey classification (DeBakey Type I, II, or III). The ascending thoracic aorta is involved in DeBakey Type I and II aortic dissections. In DeBakey Type I (ATAD), the aortic arch and descending thoracic aorta are also involved in the dissection process, therefore conventional hemiarch replacement is only considered "palliative".

Data from international registries showed the mortality of surgically treated ATAD was around 17-26% and those with mal-perfusion had even higher mortality. A significant number of patients of ATAD after conventional hemiarch replacement still have a persistent pressurized false lumen and this is related to the presence of distal anastomotic new entry (DANE).The presence of DANE leads to persistent pulsatile flow and pressurization of the false lumen in 70% of cases after hemiarch replacement.The persistently patent FL will in turn cause mal-perfusion, the need for aortic re-intervention involving the aortic arch, and, most importantly, reduced long-term survival by up to 50%.

To avoid the occurrence of DANE and downstream aortic mal-perfusion, Bozso and colleagues advocated the use of a novel Ascyrus Medical Dissection Stent (AMDS; Artivion, Atlanta, Georgia, US) hybrid prosthesis which comprises a proximal sewing collar and a distal self-expanding nitinol un-covered stent. From a prospective trial utilizing AMDS in ATAD, the Dissected Aorta Repair Through Stent Implantation (DARTS) trial, by Boszo and colleagues, the positive remodeling of the aortic arch occurred in 100% of cases with complete obliteration or thrombosis of the false lumen in 74%. In their series of 47 patients, there was no DANE after the AMDS implantation.

Work done by the principal investigator's unit is a major referral center for acute and complex aortic disease in Hong Kong, with more than 100 cases of operated aortic cases and 200 aortic referrals each year. The investigator's unit also operated on an average of 40-50 cases of ATAD each year.

The incidence of DANE in the investigator's unit is 19.5% from a retrospective reviewed of the institution's ATAD patients who received hemiarch replacement from Jan 2017 to Dec 2021. Although the incidence of DANE is lower than the reported literature, given the presence of DANE will significantly increase the risk of long-term mortality. The investigators believe a randomized control trial to compare the incidence of DANE after hemiarch replacement with or without AMDS implantation in ATAD can answer our research question and potentially be practice-changing.

Main research question is to compare the incidence of DANE after hemiarch replacement with or without AMDS implantation in acute DeBakey Type I aortic dissection.

Research methods Study Design: Single-center randomized control trial Methodology In this study, the investigators plan to prospectively recruit consecutive patients with acute DeBakey Type I aortic dissection and randomized them, after informed consent, into either the conventional hemiarch replacement group (Hemiarch-C) or the hemiarch replacement plus AMDS implantation group (Hemiarch-AMDS). The participating team will collect pre-operative, intra-operative, and post-operative clinical and radiological parameters for two groups of patients. Written informed consent, specifically allowing the use of clinical records for this randomized study, will be obtained from every patient prior to data collection. The period of data collection will be from the first recruited patient to 12 months after the last recruited patient, which will be around 36 months. Source data verification will be performed on 100% of the patients; data from all the visits that were provided in the database will be reviewed and verified against existing source documents by a dedicated research assistant. Complete DICOM image files of the CT scans will be evaluated by two independent fully qualified Radiologists. The expected patient loss rate is approximately 5% at 12 months of follow-up.

Study population Screening and randomization A computer-generated randomization sequence will be generated by the research assistant using the online randomization software. A total of 72 patients will be randomized 1:1 to one of the two treatment arms. Block randomization with block size of 8 is used to maintain good balance in each treatment group. The randomization list will be kept in a set of tamper-evident envelopes. The envelopes will be identical and sealed. The trial identifier with a sequential number will be printed on each envelope and the inside will contain the treatment allocation. Envelopes will be unsealed by the on-call surgeon to reveal the allocation treatment prior to the surgery.

Patients, with their consent, will be recruited to participate by investigators after considering the inclusion and exclusion criteria.

Blinding of the study After randomization, the recruited patient will be allocated to either AMDS or Hemiarch group. There will be no blinding of the randomization result to the recruited patients, the operating surgeons, and the clinician-in-charge.

Pre-treatment Investigations and Assessments:

1. Blood tests: complete blood count, liver and renal function tests, coagulation profile
2. Radiological imaging: CT aortogram involving the thorax and abdomen
3. ECG and/or other cardiac assessment as requested by anesthetist for general anesthesia assessment Treatment Procedures

Hemiarch-AMDS group:

Under general anesthesia and trans-esophageal echocardiogram monitoring, a median sternotomy will be performed. Patients will be put on cardiopulmonary bypass with arterial inflow from femoral artery/axillary artery/direct aortic cannulation and right atrial appendage venous two-stage cannulation. Systemic cooling to 25 Degree Celsius will commence. At a temperature of 25 Degree Celsius and thiopentone coma, the circulatory arrest will begin. The aorta will be trimmed to the level of the distal ascending or proximal arch The AMDS device will be implanted into the aortic arch and descending thoracic aorta. The distal anastomosis will be done between a vascular graft and the distal ascending aorta/aortic arch including the AMDS device sewing cuff. After the distal anastomosis is completed, visceral and cerebral systemic perfusion and rewarming will be started. The proximal ascending aorta will be anastomosed with the proximal end of the vascular graft. After de-airing and aorta will be de-clamped and the patient will be weaned from cardiopulmonary bypass and decannulated. Hemostasis and sternal closure will be done as per routine protocol.

Hemiarch-C group:

Same as above except no AMDS is implanted. The perioperative management of all recruited patients is standardized. All patients receive prophylactic antibiotics during induction and until all drains are removed in the postoperative period. All patients will have invasive blood pressure monitoring with an arterial line and intravenous antihypertensive medications aiming to control systolic blood pressure to below 140mmHg.

Sample size calculation The occurrence of DANE was estimated to be around 70% and it caused persistent false lumen perfusion, mal-perfusion, early mortality, and decreased long-term survival. From a prospective trial by Moon and colleagues, the positive remodeling of the aortic arch occurred in 100% of cases with complete obliteration or thrombosis of the false lumen in 74%. In their series of 47 patients, there was no DANE after the AMDS implantation. Our own unpublished cohort of 167 cases revealed the occurrence of DANE in 19.5% after our hemiarch procedures. Based on a previous report and our own cohort of DANE rate of 19.5% and 70% respectively, and assumed DANE rate of 0% after AMDS, 36 patients need to be recruited for each arm (a total of 72 patients) in order to demonstrate a statistically significant difference with an 80% power at the 0.05 level of 1-sided significant difference between Hemiarch-AMDS and Hemiarch-C by a superiority time-to-event study design.

Data analysis Statistical analysis will be performed using SPSS version 28.0.0.0 (IBM, NewYork, USA) on an intention-to-treat basis. The primary analysis set for statistical reporting will be the ITT population with no replacement of missing data planned in the statistical analysis to provide unbiased results. Missing data will be checked, and the imputation of the missing data will be used to preserve statistical power. The investigators will use the log-rank test to compare the time from randomization to the endpoints of occurrence of DANE. A Cox proportional-hazards model to estimate the hazard ratio and 95% confidence intervals. The investigators will use Schoenfeld residual test to verify the assumption of proportional hazards in the Cox analysis, to fulfill the endpoint of the occurrence of DANE. Secondary endpoints will be compared between groups with a chi-square test for difference in proportions with student's t-test and a Mann-Whitney U test for parametric and non-parametric data, respectively. All tests of significance were two-tailed, and a P value of 0.05 or less will be considered to indicate statistical significance for the primary endpoint. Percentages will be calculated on the number of non-missing observations. When applicable, bilateral asymptotic or exact confidence intervals (CIs) for binomial distributions will be calculated at the 95% level (unadjusted 95% CI). For analysis of data where the outcome variable is the time until the occurrence of an event of interest (for example, death, myocardial infarction etc.), the non-parametric estimator of these survival functions will be presented using the Kaplan-Meier method, together with a graphical presentation.

The investigator's unit operate on an average of 40-50 cases of acute aortic dissection each year. Assuming DeBakey Type I (ATAD) constitutes around 87% of all acute aortic dissection and acceptance of study by patients of 90%. It is therefore expected that recruitment can be completed in about 24 months. The last recruited patient will be observed for at least 12 months after the procedure. Hence, the total period of study including follow-up is 3 years, which is also the funding period for the grant application. After completion of the funding period, the recruited patients will be followed up to 2 years with interval investigations with CT scans to assess the aortic remodeling of both groups.

All clinical data will be collected in the principal investigator's center by a dedicated research assistant. Continuous clinical data monitoring and interim and final analysis will be performed by the principal investigator and co-investigators with the help of a research assistant.

Ethical consideration This study shall be conducted in accordance with the ethical principles in the Declaration of Helsinki. This protocol is approved by the Joint Chinese University of Hong Kong and New Territories East Cluster Clinical Research Ethics Committees (CREC:2023.075-T)). Written informed consent, specifically allowing the use of clinical records for study purposes, will be obtained from every patient prior to data collection.

Patients can withdraw from the study without any prejudice at any time during the study. Data will be kept confidential in secure offices of the Department of Surgery for seven years.

Potential risks of the study Acute aortic dissection is a life-threatening emergency condition with mortality of around 17-26% from the world registries. In the principal investigator unit, from a retrospective record review of 2017-2021, the investigator's center has 167 Acute aortic dissection. Among this cohort, there was 87.1% of patients with DeBakey Type I (ATAD). Our operative mortality for ATAD is 4.3%. The incidence of DANE in our patients is 19.5%. According to the DARTS trial, the placement of AMDS device increases circulatory arrest time by an average of 3 minutes with 100% technical success rate. The implantation of AMDS is simple and much more generalizable than the complicated TARFET. The investigators do not anticipate there will be any increase in mortality or morbidity with AMDS implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient´s age is between 18 and 80 years.
2. Patient is willing and able to give informed consent.
3. Patient has acute DeBakey Type I and requires repair or replacement of damaged or diseased vessels of the ascending aorta.
4. Patient not in coma/irreversible end organ failure/cardiac massage for resuscitation, at the time of consent.

Exclusion Criteria:

1. Patient has aortic arch diameter of more than 4.5 cm
2. Patient has known connective tissue disease or genetically linked aortopathy
3. Patient has entry tear more than 2 cm over aortic arch
4. Patient with DeBakey Type II aortic dissection
5. Patient has co-morbidity (i.e. active malignancy (progressive, stable or partial remission)) causing expected survival to be less than 2 years.
6. Patient has any other medical, social, or psychological problems, that in the opinion of the investigator, preclude the patient from participating in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of DANE | At Discharge(0-14days), 30-day, 3-6 month, 12 month
  The presence of Distal Anastomosis New Entry (DANE) diagnosed by Computed Tomography in post-operative imaging within the 12-month follow-up period

SECONDARY OUTCOMES:
All-cause mortality of the patients | At discharge(0-14days), 30-day, 3-6 month, 12 month
  Rate of death in the whole cohort
Percentage of patient with aortic-related mortality | At Discharge(0-14days), 30-day, 3-6 month, 12 month
  Percentage of patient that die from aortic related event
Percentage of patients with Major Adverse Events | At Discharge(0-14days), 30-day, 3-6 month, 12 month
  Rate of patients who are free from the following Major Adverse Events (MAEs) (new permanent disabling stroke), new permanent (> 30 days) paraplegia or paraparesis, reintervention (excluding reoperation for bleeding or planned or unplanned additional intervention), visceral mal-perfusion, limb(s) ischemia
Percentage of patients requiring additional aortic intervention | At Discharge(0-14days), 30-day, 3-6 month, 12 month
  Rate of patients with aortic rupture and additional intervention (planned / unplanned)
Percentage of patients with Renal failure | At Discharge(0-14days), 30-day, 3-6 month, 12 month
  Renal failure requiring permanent (> 90 days) dialysis or hemofiltration in a patient with a normal pre-procedure serum creatinine level
Percentage of patients with radiological head and neck vessels patency | At Discharge(0-14days), 30-day, 3-6 month, 12 month
  Radiological patency in supra-aortic head vessels (0 - 30 %, >30 % - 50 %, > 50 % - 70%, > 70%) (kink-, suture line-, dissection-related, other)
Percentage of patient with failure of AMDS | At Discharge(0-14days), 30-day, 3-6 month, 12 month
  Failure of the integrity of the AMDS
Percentage of patients with radiological true and false lumen status of the aortic arch and descending thoracic aorta | At Discharge(0-14days), 30-day, 3-6 month, 12 month
  Radiological findings of the true lumen, false lumen thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
Anonymized clinical and radiological outcome data will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available when we complete our analysis and for a 12-month period
Access Criteria: Approval needs to be sought from the Principal Investigator

REFERENCES:
- [Background] Hagan PG, Nienaber CA, Isselbacher EM, Bruckman D, Karavite DJ, Russman PL, Evangelista A, Fattori R, Suzuki T, Oh JK, Moore AG, Malouf JF, Pape LA, Gaca C, Sechtem U, Lenferink S, Deutsch HJ, Diedrichs H, Marcos y Robles J, Llovet A, Gilon D, Das SK, Armstrong WF, Deeb GM, Eagle KA. The International Registry of Acute Aortic Dissection (IRAD): new insights into an old disease. JAMA. 2000 Feb 16;283(7):897-903. doi: 10.1001/jama.283.7.897. PMID 10685714
- [Background] Czerny M, Schoenhoff F, Etz C, Englberger L, Khaladj N, Zierer A, Weigang E, Hoffmann I, Blettner M, Carrel TP. The Impact of Pre-Operative Malperfusion on Outcome in Acute Type A Aortic Dissection: Results From the GERAADA Registry. J Am Coll Cardiol. 2015 Jun 23;65(24):2628-2635. doi: 10.1016/j.jacc.2015.04.030. PMID 26088302
- [Background] Bozso SJ, Nagendran J, Chu MWA, Kiaii B, El-Hamamsy I, Ouzounian M, Kempfert J, Starck C, Moon MC. Midterm Outcomes of the Dissected Aorta Repair Through Stent Implantation Trial. Ann Thorac Surg. 2021 Feb;111(2):463-470. doi: 10.1016/j.athoracsur.2020.05.090. Epub 2020 Jul 13. PMID 32673661
- [Background] Rylski B, Hahn N, Beyersdorf F, Kondov S, Wolkewitz M, Blanke P, Plonek T, Czerny M, Siepe M. Fate of the dissected aortic arch after ascending replacement in type A aortic dissectiondagger. Eur J Cardiothorac Surg. 2017 Jun 1;51(6):1127-1134. doi: 10.1093/ejcts/ezx062. PMID 28369453
- [Background] Evangelista A, Salas A, Ribera A, Ferreira-Gonzalez I, Cuellar H, Pineda V, Gonzalez-Alujas T, Bijnens B, Permanyer-Miralda G, Garcia-Dorado D. Long-term outcome of aortic dissection with patent false lumen: predictive role of entry tear size and location. Circulation. 2012 Jun 26;125(25):3133-41. doi: 10.1161/CIRCULATIONAHA.111.090266. Epub 2012 May 21. PMID 22615344
- [Background] Kobuch R, Hilker M, Rupprecht L, Hirt S, Keyser A, Puehler T, Amman M, Zink W, Schmid C. Late reoperations after repaired acute type A aortic dissection. J Thorac Cardiovasc Surg. 2012 Aug;144(2):300-7. doi: 10.1016/j.jtcvs.2011.08.052. Epub 2011 Nov 12. PMID 22078710
- [Background] Halstead JC, Meier M, Etz C, Spielvogel D, Bodian C, Wurm M, Shahani R, Griepp RB. The fate of the distal aorta after repair of acute type A aortic dissection. J Thorac Cardiovasc Surg. 2007 Jan;133(1):127-35. doi: 10.1016/j.jtcvs.2006.07.043. Epub 2006 Dec 4. PMID 17198797
- [Background] Kimura N, Itoh S, Yuri K, Adachi K, Matsumoto H, Yamaguchi A, Adachi H. Reoperation for enlargement of the distal aorta after initial surgery for acute type A aortic dissection. J Thorac Cardiovasc Surg. 2015 Feb;149(2 Suppl):S91-8.e1. doi: 10.1016/j.jtcvs.2014.08.008. Epub 2014 Aug 13. PMID 25224548
- [Background] Shrestha M, Pichlmaier M, Martens A, Hagl C, Khaladj N, Haverich A. Total aortic arch replacement with a novel four-branched frozen elephant trunk graft: first-in-man results. Eur J Cardiothorac Surg. 2013 Feb;43(2):406-10. doi: 10.1093/ejcts/ezs296. Epub 2012 May 31. PMID 22653445
- [Background] Shrestha M, Haverich A, Martens A. Total aortic arch replacement with the frozen elephant trunk procedure in acute DeBakey type I aortic dissections. Eur J Cardiothorac Surg. 2017 Jan;51(suppl 1):i29-i34. doi: 10.1093/ejcts/ezw341. PMID 28108566
- [Background] Dohle DS, Tsagakis K, Janosi RA, Benedik J, Kuhl H, Penkova L, Stebner F, Wendt D, Jakob H. Aortic remodelling in aortic dissection after frozen elephant trunkdagger. Eur J Cardiothorac Surg. 2016 Jan;49(1):111-7. doi: 10.1093/ejcts/ezv045. Epub 2015 Feb 24. PMID 25715431
- [Background] Tsagakis K, Dohle DS, Wendt D, Wiese W, Benedik J, Lieder H, Thielmann M, Jakob H. Left subclavian artery rerouting and selective perfusion management in frozen elephant trunk surgery. Minim Invasive Ther Allied Technol. 2015;24(5):311-6. doi: 10.3109/13645706.2015.1069358. PMID 26358834
- [Background] Bozso SJ, Nagendran J, Chu MWA, Kiaii B, El-Hamamsy I, Ouzounian M, Kempfert J, Starck C, Shahriari A, Moon MC. Single-Stage Management of Dynamic Malperfusion Using a Novel Arch Remodeling Hybrid Graft. Ann Thorac Surg. 2019 Dec;108(6):1768-1775. doi: 10.1016/j.athoracsur.2019.04.121. Epub 2019 Jun 27. PMID 31254509
- [Background] Bozso SJ, Nagendran J, MacArthur RGG, Chu MWA, Kiaii B, El-Hamamsy I, Cartier R, Shahriari A, Moon MC. Dissected Aorta Repair Through Stent Implantation trial: Canadian results. J Thorac Cardiovasc Surg. 2019 May;157(5):1763-1771. doi: 10.1016/j.jtcvs.2018.09.120. Epub 2018 Oct 26. PMID 30501947
- [Background] Montagner M, Kofler M, Heck R, Buz S, Starck C, Kurz S, Falk V, Kempfert J. Initial experience with the new type A arch dissection stent: restoration of supra-aortic vessel perfusion. Interact Cardiovasc Thorac Surg. 2021 Jul 26;33(2):276-283. doi: 10.1093/icvts/ivab085. PMID 34010408
- [Background] Mehdiani A, Sugimura Y, Wollgarten L, Immohr MB, Bauer S, Schelzig H, Wagenhauser MU, Antoch G, Lichtenberg A, Akhyari P. Early Results of a Novel Hybrid Prosthesis for Treatment of Acute Aortic Dissection Type A With Distal Anastomosis Line Beyond Aortic Arch Zone Zero. Front Cardiovasc Med. 2022 Jul 14;9:892516. doi: 10.3389/fcvm.2022.892516. eCollection 2022. PMID 35911517
- [Background] Wong RH, Baghai M, Yu SC, Underwood MJ. Aortic arch/elephant trunk procedure with Sienna(TM) graft and endovascular stenting of thoraco-abdominal aorta for treatment of complex chronic dissection. Ann Cardiothorac Surg. 2013 May;2(3):358-61. doi: 10.3978/j.issn.2225-319X.2013.05.03. PMID 23977606
- [Background] Wong RH, Yu SC, Lau RW, Ng CS, Hui JW, Wan IY, Wan S, Ho AM, Underwood MJ. Delayed stent deformity and fracture of Djumbodis dissection system. Ann Thorac Surg. 2014 Jan;97(1):e17-20. doi: 10.1016/j.athoracsur.2013.07.127. PMID 24384216
- [Background] Wong RH, Ho JY, Underwood MJ. Multimodality imaging assessment for Thoraflex hybrid total arch replacement. Asian Cardiovasc Thorac Ann. 2016 Jun;24(5):496-501. doi: 10.1177/0218492316643844. Epub 2016 Apr 11. PMID 27072867
- [Background] Ho JYK, Chow SCY, Kwok MWT, Fujikawa T, Wong RHL. Total Aortic Arch Replacement and Frozen Elephant Trunk. Semin Thorac Cardiovasc Surg. 2021 Autumn;33(3):656-662. doi: 10.1053/j.semtcvs.2020.11.016. Epub 2020 Nov 9. PMID 33181309
- [Background] Ho JYK, Bashir M, Jakob H, Wong RHL. Management of left subclavian artery in total arch replacement and frozen elephant trunk procedure. JTCVS Tech. 2021 Mar 29;7:36-40. doi: 10.1016/j.xjtc.2021.03.020. eCollection 2021 Jun. No abstract available. PMID 34318200
- See also: Block randomization — https://www.sealedenvelope.com/simple-randomiser/v1/lists
- See also: Sample size calculator — https://clincalc.com/stats/SampleSize.aspx
- See also: Video 1 — https://youtu.be/Nbl37-Ca2hM
- See also: Centre for Health Protection, Vital Statistics, Death Rates by Leading Causes of Death 1981-2000 — http://www.chp.gov.hk/en/data/4/10/27/115.html
- See also: Hospital Authority Statistical Report 2009-2010, Page 28, Table 1.1 — http://www.ha.org.hk/upload/publication_15/321.pdf
- See also: Hospital Authority Statistical Report 2011-2012, Page 30, Table 1.2 — http://www.ha.org.hk/upload/publication_15/471.pdf
- See also: Wong RH, Ho JY, Bashir M, Jakob H. First-in-man implantation of Evita Open Neo in Hong Kong. CTSNet 2020. — https://doi.org/10.25373/ctsnet.13373762.v1